CLINICAL TRIAL: NCT06156605
Title: Looking Beyond the Immediate Effects of Lumbar Spinal Manipulation Using Pain Pressure Threshold in Asymptomatic Individuals
Acronym: LumbarPPTUMary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mary (Other)
Responsible Party: Principal Investigator, Matthew Schumacher, Dr. Schumacher, PT, DPT, OCS, FAAOMPT, University of Mary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMary1234
Record Dates: First submitted 2023-11-25; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Lumbar Spine Injury; Pain
MeSH Terms: conditions — Spinal Injuries; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sidelying lumbar manipulation (Experimental): Right sided lumbar manipulation
  Interventions: Procedure: Sidelying lumbar manipulation
- Sham ultrasound (Active Comparator): Sham (non-therapeutic settings) ultrasound at the right PSIS
  Interventions: Procedure: Sidelying lumbar manipulation

INTERVENTIONS:
Procedure: Sidelying lumbar manipulation — R sided lumbar manipulation

SUMMARY:
The goal of this clinical trial is to test in the effects of pain pressure threshold (PPT) looking out to 30 minutes in the lumbar spine. The main question[s] it aims to answer are:

• Is there a difference between PPT from baseline, immediately after, or 30 minutes after compared to sham ultrasound control group? Participants will be exposed to sham ultrasound or sidelying lumbar manipulation with between groups and within group comparisons of PPT at the posterior superior iliac spine up to 30 minutes following the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic individuals between the ages of 18-50

Exclusion Criteria:

* Current low back pain (LBP)
* A history of low back pain LBP within the last three months
* Previous spinal surgery
* Rheumatological condition or neurological symptoms or conditions
* Recent ingestion of pain-relieving medications within the last 24 hours
* A lumbar manipulation within three days prior to the exam
* Exhibited any contraindications to manipulation
* Positive findings during screening precautions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold | Baseline, Immediately after, 30 minutes after
  PPT at the right PSIS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mary, Bismarck, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schumacher MR, Swanson C, Wolff S, Orteza R, Aguilar R. Exploring the immediate and short-term effect of lumbar spinal manipulation on pressure pain threshold: a randomized controlled trial of healthy participants. Chiropr Man Therap. 2024 May 29;32(1):19. doi: 10.1186/s12998-024-00540-5. PMID 38811985